CLINICAL TRIAL: NCT00979290
Title: Comparison of Adverse Reactions and Efficiency of Fixed-dose Combination Chemotherapy and Separate Formulations for Pulmonary Tuberculosis
Brief Title: Adverse Reactions and Efficacy of Fixed-dose Combination Anti-tuberculosis (TB) Drugs
Status: Completed | Type: Observational
Sponsor: E-DA Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: J120114933
Record Dates: First submitted 2009-09-14; First posted 2009-09-17 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Tuberculosis
Keywords: Fix-dose combination anti-TB drug; adverse effect; efficiency
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Separate anti-TB drugs
- Fix-dosed combination anti-TB drugs

SUMMARY:
The fixed-dose combinations (FDC) with two or more antituberculous drugs in one capsule or tablet are available to prevent the development of drug resistance. However, the fixed-dose combination regimen is not consistent with the dosages that are usually given. The present available FDC chemotherapy (Rifater) for pulmonary tuberculosis that is used in Taiwan has a higher ratio of isoniazid to rifampin and pyrazinamide. The higher risk of drug toxicity and adverse reactions when using fixed-dose combinations regimen should be considered. The aim of the present study is to compare the toxicity between using FDC regimen (Rifater/Rifinah) in Taiwan and single drugs in the treatment of newly diagnosed pulmonary tuberculosis. The investigators also evaluate the efficacy of two regimens and determine the incidence of discontinuation of TB drugs and the predisposed factors between two regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed pulmonary TB and extrapulmonary TB patients
2. No previous anti-TB drugs treatment
3. Age≥18years old

Exclusion Criteria:

1. Expected life < 6months
2. Baseline AST/ALT > 3x upper limit of normal (ULN)
3. Age <18years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed TB patients in E-DA hospital
Sampling Method: Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To compare the frequency of occurrence of adverse reactions between using FDC and single drugs in pulmonary tuberculosis treatment | two year

SECONDARY OUTCOMES:
To compare the efficacy of anti-TB treatment between using FDC and single drugs | two year

CONTACTS AND LOCATIONS:
Locations (1):
- E-DA hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Wu JT, Chiu CT, Wei YF, Lai YF. Comparison of the safety and efficacy of a fixed-dose combination regimen and separate formulations for pulmonary tuberculosis treatment. Clinics (Sao Paulo). 2015 Jun;70(6):429-34. doi: 10.6061/clinics/2015(06)08. Epub 2015 Jun 1. PMID 26106962